CLINICAL TRIAL: NCT05240625
Title: Clinical Efficacy Evaluation of a Computer-aided Colonoscopy as Compared With the Standard Colonoscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Changhua Christian Hospital (Other); Shin Kong Hospital (Unknown); Fu Jen Catholic University Hospital (Other); aetherAI Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 202112052DIPC
Record Dates: First submitted 2022-02-13; First posted 2022-02-15 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-01

CONDITIONS: Colon Adenoma; Colorectal Cancer
Keywords: Computer-aided colonoscopy; Artificial intelligence; Colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Delivery Systems; Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject and the pathologist who performs the histopathological review will be blinded to the received procedure, while the operator for colonoscopy will not be blinded to the study arm assigned to the subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-aided colonoscopy (Experimental): The subject will receive the standard colonoscopy procedure simultaneously with a computer-aided detection (CADe) analysis software designed to automatically detect and highlight potential polyps on colonoscopy images in a real-time manner during colonoscopy procedures.
  Interventions: Device: "aetherAI" Computer-aided Polyp Detection (CADe) Systems for Colonoscopy; Procedure: Standard colonoscopy
- Standard colonoscopy (Active Comparator): The subject will receive the standard colonoscopy procedure.
  Interventions: Procedure: Standard colonoscopy

INTERVENTIONS:
Device: "aetherAI" Computer-aided Polyp Detection (CADe) Systems for Colonoscopy — The investigational medical device is intended to automatically detect potential polyps via colonoscopy in real-time during colonoscopy examinations.
  The subject device contains an artificial intelligence/machine learning (AI/ML) advanced algorithm to aid the endoscopists in detection of colonic mucosal lesions and the detected polyps will be highlighted to the endoscopists during the real-time colonoscopy procedures.
  Arms: Computer-aided colonoscopy
Procedure: Standard colonoscopy — Standard colonoscopy procedure.

SUMMARY:
Colonoscopy is clinically used as the gold standard for detection of colorectal cancer (CRC) and removal of adenomatous polyps of the colon and rectum. Evidence has shown that CRC could be prevented by colonoscopic removal of adenomatous polyps. Despite the success of colonoscopy in reducing cancer-related deaths, there exists a disappointing level of adenomas missed at colonoscopy. In recent years, emerging artificial intelligence (AI) and computer-aided detection (CADe) technology has been shown to improve ADR. Based on a meta-analysis, ADR was demonstrated to be significantly higher in the CADe groups than in the standard colonoscopy groups, representing a relative risk of 25.2%.

In this study, performance of colonoscopy with or without aid of CADe will be compared in terms of quality indicators. The adenoma detection rate (ADR), which is the proportion of average-risk patients undergoing screening colonoscopy in whom an adenoma is found, is regarded as a robust measure of colonoscopy performance quality that correlates with subsequent cancer risk. Thus, ADR is taken as the primary outcome of this study. The target population includes individuals who are undergoing screening, diagnostic, or surveillance colonoscopy.

DETAILED DESCRIPTION:
This multiple-site study aims to evaluate whether a computer-aided detection (CADe) device can assist in adenoma detection rate (ADR) when compared with the current standard-of-care procedure. The subject CADe device used in this study contains an artificial intelligence/machine learning (AI/ML) advanced algorithm to aid the endoscopists in detection of colonic mucosal lesions and the detected polyps will be highlighted to the endoscopists during the real-time colonoscopy procedures. This study plans to enroll subjects aged ≥ 40 years and < 80 years, who are scheduled for screening or diagnostic colonoscopy for colorectal cancer (CRC) or surveillance colonoscopy for post-polypectomy follow-up. After being evaluated with the inclusion and exclusion criteria, eligible subjects will be randomized in a 1:1 ratio to receive either the computer-aided colonoscopy (CC) or the standard colonoscopy(SC). Randomization will be stratified by gender, age, and colonoscopy indication (screening, diagnostic, or surveillance) of subjects. The resected polyps will be submitted for histologic examination by one expert pathologist at each site. If any uncertainty or doubt exists, an expert in gastrointestinal pathology will serve as the adjudicator to perform a second review and make the final decision. All of the pathologists (including the final adjudicator) who will perform the histopathologic examinations and produce the pathology assessment will be blinded to the assigned study arm of the specimens. The pathology reports of the subjects will be kept securely at each site as the source data.

The primary endpoint is the ADR of the CC as compared with that of the SC. The ADR is defined as the percentage of subjects undergoing a complete colonoscopy, who have at least one histologically confirmed adenoma detected and removed. In addition, the following secondary endpoints will also be evaluated, including: Polyp detection rate (PDR), Adenomas per colonoscopy (APC), Polyps per colonoscopy (PPC), Non-neoplastic polypectomy rate (NNPR), Non-neoplastic polypectomy (NNP), Sessile serrated lesions per colonoscopy (SPC), Advanced adenomas per colonoscopy (AAPC), and withdrawal time.

Signed written informed consent forms will be obtained from all participating subjects before enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have given signed informed consent form
* Informed consensus has been obtained that endoscopic resection should be performed if a lesion is found
* Subjects who are scheduled for screening or diagnostic colonoscopy for colorectal cancer (CRC) or surveillance colonoscopy for post-polypectomy follow-up

Exclusion Criteria:

* Subjects with any of the following prior history or current conditions:

  1. Contraindications to colonoscopy
  2. Inflammatory bowel disease (IBD)
  3. Colorectal cancer (CRC)
  4. Familial adenomatous polyposis (FAP)
  5. Colonic stenosis
  6. Severe organ failure (cirrhosis of Child C, heart failure of ACC / AHA stage D)
  7. Active gastrointestinal (GI) Bleeding
  8. Pregnancy
  9. Prior colorectal surgery, including colonic or rectal resection (except for appendectomy, surgery on the anus, and polypectomy)
  10. Undergo colonoscopy within 3 years
* Subjects with any of the following conditions per the investigator's judgement:

  1. High suspicion of IBD, CRC, and FAP.
  2. High risk of bleeding after endoscopic treatment, and difficult management of anticoagulation or antiplatelet medication.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 week (after the colonoscopy procedure, when pathology report is released)
  The percentage of subjects undergoing a complete colonoscopy, who have at least one histologically confirmed adenoma detected and removed.

SECONDARY OUTCOMES:
Polyp detection rate (PDR) | 1 day(right after the colonoscopy procedure)
  Percentage of subjects undergoing a complete colonoscopy who have at least one polyp detected.
Adenomas per colonoscopy (APC) | 1 week (after the colonoscopy procedure, when pathology report is released)
  Number of adenomas per colonoscopy, calculated by dividing the total number of adenomas detected by the total number of colonoscopies.
Polyps per colonoscopy (PPC) | 1 day(right after the colonoscopy procedure)
  Number of polyps of any kind (i.e., adenoma, sessile serrated polyp, hyperplastic polyp, or non-neoplastic polyp) per colonoscopy, calculated by dividing the total number of polyps detected by the total number of colonoscopies.
Non-neoplastic polypectomy rate (NNPR) | 1 week (after the colonoscopy procedure, when pathology report is released)
  Percentage of subjects with at least one non-neoplastic polypectomy at the time of colonoscopy.
Sessile serrated lesions per colonoscopy (SPC) | 1 week (after the colonoscopy procedure, when pathology report is released)
  Number of sessile serrated lesions (SSLs) per colonoscopy, calculated by dividing the total number of sessile serrated lesions detected by the total number of colonoscopies.
Advanced adenomas per colonoscopy (AAPC) | 1 week (after the colonoscopy procedure, when pathology report is released)
  Number of advanced adenomas per colonoscopy, calculated by dividing the total number of advanced adenomas detected by the total number of colonoscopies.
Withdrawal time | 1 day(right after the colonoscopy procedure)
  The time spent in inspecting the colonic mucosa as the endoscope is withdrawn during a colonoscopy, excluding procedure time

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Not shareable due to local IRB considerations.